CLINICAL TRIAL: NCT03498924
Title: Prospective Identification and Characterization of Endometrial Cancer With Specific Tumor Markers in Serum and Endometrial Tissue Samples
Brief Title: Identification and Characterization of Endometrial Cancer With Specific Tumor Markers in Serum and Endometrial Tissue
Status: Completed | Type: Observational
Sponsor: Fundación Investigación Sanitaria en León (Other)
Responsible Party: Principal Investigator, Tatiana Cuesta-Guardiola, Principal investigator, Fundación Investigación Sanitaria en León
Other Study IDs: STUDY17104
Record Dates: First submitted 2018-02-23; First posted 2018-04-17 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Endometrial Neoplasm Malignant
Keywords: tumor marker; HE4; CA125; staging; diagnosis; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and endometrial tissue sample of every patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASES: Patients with endometrial cancer
  Interventions: Diagnostic Test: Measure of biomarkers in serum and endometrial tissue
- CONTROLS: Matched controls without neoplasm disease
  Interventions: Diagnostic Test: Measure of biomarkers in serum and endometrial tissue

INTERVENTIONS:
Diagnostic Test: Measure of biomarkers in serum and endometrial tissue — Blood sample and endometrial sample

SUMMARY:
Endometrial cancer is the most common malignant tumor of the female genital tract in our means. The diagnosis is made by endometrial biopsy sampling with anatomopathological analysis which pinpoints the cell line and the level of cell differentiation. Its treatment is surgical with adjuvant treatment (chemotherapy or radiotherapy) besides, depending on the staging. Thus far, in the first diagnosis it is only request the tumor marker CA125 in serum, but there are studies that identify the HE4 protein in blood as a feasible marker for endometrial cancer. Furthermore, the staging changes the surgical and the adjuvant treatment: in its early stages, surgery is based on hysterectomy and double adnexectomy, however, in later stages it is necessary to add pelvic and paraaortic lymphadenectomy with the associated comorbidity. This makes extremely important that the preoperative diagnosis is accurate. The aim of this study is to identify and characterize the HE4, Ki67, p53 and other potential biomarkers in endometrial tissue in order to diagnose patients with disease only with a biopsy. Moreover, the investigators are searching for connections among these markers and prognostic factors such as grade of cell differentiation, cell line, lymphatic affectation, tumor stage or even features as survival or disease free survival.

DETAILED DESCRIPTION:
List of abbreviations:

* HE4: Human Epididymis Protein 4
* CA125: Carbohydrate Antigen 125
* Ki67: antigen KI67
* EC: Endometrial Cancer
* CT: Computed Tomography
* NMR: Nuclear Magnetic Resonance
* FIGO: International Federation of Gynecology and Obstetrics

The purpose of this study is:

* The proportion of positive H-score of HE4, as quantified in endometrial tissue. It is significantly higher in patients with endometrial cancer than in non-EC patients.
* Percentage of HE4, CA125 and other markers positives in cases and controls.
* Concentration of HE4 in tissue, as measured by H-score, correlates linearly with HE4 concentration in serum, as measured in terms of ppmol/l.
* Differences in serum CA125 levels between cases and controls.
* Quantification of tissue tumor markers of EC patients, per disease stages.
* Relation of the immunohistochemistry intensity with survival and disease-free survival times.
* Analysis of other risk factors adjusting for known variables like age, menopausal status, hypertension, diabetes or obesity.
* Feasibility of the technique.

Steps in the study:

1. Patients enter the study when a diagnosis of endometrial cancer is done. As it is ordinary in the clinical practice the diagnosis is made with an endometrial tissue sample taken in the office which is afterwards studied by a pathologist, who makes the final diagnosis.
2. Patients undergo the regular preoperative study with pelvic ultrasound, CT and/or NMR for the extension study, blood tests and the preanaesthetic consultation. As it is registered in the protocol of Endometrial Cancer Treatment.
3. Then a matched control is selected from the group of patients that are going to be hysterectomized for other non-malignant reasons (abdominal way, vaginal, or laparoscopic way). Variables considered for matching are: age (variability of five years), pre or postmenopausal status, hypertension, obesity and diabetes.
4. Every patient then is asked for accept and sign the informed consent. The next step is to prepare the patient for the surgery. In this moment the serum sample is taken. Subsequently the surgery will be performed.
5. Then the anatomopathological study is conducted over the preoperative tissue sample. HE4 marker in endometrial tissue is defined by H-Score while Ki67 and p53 are defined as usual. Although Ki67 is matched in > or <25% of expression instead of 14% as it is made in breast cancer tissue samples.
6. After discharge, the patient will be follow-up for two years in order to register the evolution of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Of legal age (≥ 18 years)
* Wish to participate in the research study and sign consent forms voluntarily
* Patients diagnosed of endometrial cancer derived to hysterectomy

Exclusion Criteria:

* Patients that underwent surgery for other malignant pathologies, whether for ovarian carcinoma, cervical carcinoma or uterine sarcoma.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Every patient who is treated in Hospital de Leon of endometrial disease between August 2017 and the end of the recruitment
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
The proportion of positive H-score of HE4. | Two years
  HE4 quantified in endometrial tissue is significantly higher in patients with endometrial cancer than in non-EC patients

SECONDARY OUTCOMES:
Concentration of HE4 in tissue correlates linearly with HE4 in serum. | Two years
  Comparison of tissue H-score with ppmol/L in serum
Difference in preoperative serum CA125 levels in cases and controls. | Two years
  Measured in terms of U/mL
Difference in preoperative serum HE4 levels in cases and controls. | Two years
  Measured in terms of ppmol/L
Disease stages | Two years
  FIGO stages: postsurgical classification drawn up to define the extent of spread of genital cancer
Tissue tumor marker HE4 | Two years
  H-score determination: Immunohistochemistry results can be evaluated by a semiquantitative approach used to assign an H-score (or "histo" score) to tumor samples. Cytoplasmic staining will be graded for intensity (0-negative, 1-weak, 2-moderate and 3-strong) and the percentage of positive cells was scored as 0 (0%), 1 (1-10%), 2 (11-50%) and 3 (51-100%).
  Single scale with scores 0-9 will be obtained by multiplying the intensity and the percentage staining score, and a total score will be calculated by grouping score 0 in total score 0, 1-3 in total score 1, 4-6 in total score 2 and 7-9 in total score 3.
  The assumption is that as higher is the score the level of cell differentiation would be minor.
Relation of the immunohistochemistry intensity in H-score with overall survival | Through study completion, an average of 2 years
  HE4 biomarker measured with H-score in endometrial tissue, explained in outcome 5, in relation to length of time of survival
Relation of the immunohistochemistry intensity in H-score with disease-free survival | Through study completion, an average of 2 years
  HE4 biomarker measured with H-score in endometrial tissue, explained in outcome 5, in relation to length of time after primary treatment that the patient survives without any signs or symptoms of that cancer.
Analysis of outcomes in relation to age | Two years
  Age of patients is one of the known risk factors for EC, we are going to analysis the results of the study with this variable. As elder the relative risk is higher though there is no accurate cut-off point.
Analysis of outcomes in relation to menopausal status | Two years
  Menopausal status is determined by questionnaire during the preoperative consultant. It is another risk factor for EC, the postmenopausal status has higher relative risk than premenopausal status.
Analysis of outcomes in relation to hypertension | Two years
  Hypertension is diagnosed previously to surgery as Blood Pressure over 140/90 mm Hg in several measures. There is a known high relative risk of EC in patients diagnosed with hypertension.
Analysis of outcomes in relation to diabetes | Two years
  Diabetes is a disease previously diagnosed by high glucose levels in blood. There is a known high relative risk of EC in patients diagnosed with diabetes.
Analysis of outcomes in relation to obesity | Two years
  Obesity is defined as BMI >27 kg/m2. There is a known high relative risk of EC in patients diagnosed with obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Cuesta-Guardiola, Medicine, Principal Investigator — Hospital de Leon
Locations (1):
- Tatiana Cuesta-Guardiola, León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Result] Creasman WT, Morrow CP, Bundy BN, Homesley HD, Graham JE, Heller PB. Surgical pathologic spread patterns of endometrial cancer. A Gynecologic Oncology Group Study. Cancer. 1987 Oct 15;60(8 Suppl):2035-41. doi: 10.1002/1097-0142(19901015)60:8+3.0.co;2-8. PMID 3652025
- [Result] Li X, Gao Y, Tan M, Zhuang H, Gao J, Hu Z, Wang H, Zhu L, Liu J, Lin B. Expression of HE4 in Endometrial Cancer and Its Clinical Significance. Biomed Res Int. 2015;2015:437468. doi: 10.1155/2015/437468. Epub 2015 Oct 11. PMID 26539494
- [Result] Bignotti E, Ragnoli M, Zanotti L, Calza S, Falchetti M, Lonardi S, Bergamelli S, Bandiera E, Tassi RA, Romani C, Todeschini P, Odicino FE, Facchetti F, Pecorelli S, Ravaggi A. Diagnostic and prognostic impact of serum HE4 detection in endometrial carcinoma patients. Br J Cancer. 2011 Apr 26;104(9):1418-25. doi: 10.1038/bjc.2011.109. Epub 2011 Apr 5. PMID 21468050
- See also: Cancer Research UK. Uterine Cancer Statistics. — http://www.cancerresearchuk.org/health-professional/cancer-statistics/statistics-by-cancer-type/uterine-cancer#heading-Zero.
- See also: Group, U.S. Cancer Statistics Working. United States Cancer Statistics: 1999-2014 Incidence and Mortality Web-based Report. — http://www.cdc.gov/uscs.